CLINICAL TRIAL: NCT02253511
Title: A Prospective Randomized Control Study of Cidan Capsule Combined With Transcatheter Arterial Chemoembolization in Hepatocellular Carcinoma
Brief Title: A Prospective Control Study of Cidan Capsule Combined With TACE in Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zheng Donghai (Other Government)
Responsible Party: Sponsor-Investigator, Zheng Donghai, Vice-President of Beijing Weida Cancer Hospital of Chinese Traditional Medical Sciences, Beijing Weida Cancer Hospital of Chinese Traditional Medical Sciences
Organization: Beijing Weida Cancer Hospital of Chinese Traditional Medical Sciences (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-2014; NST-CD (Other Grant/Funding Number: Key Project of NST, 2013ZX09104-006)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepotectomy; Recurrence-free survival; Overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cidan capsule (Experimental): Patients who undergone operation and TACE were administered 1.35 g cidan capsules (Weida Pharmaceutical Co., Ltd., Beijing, China) three times a day for 3 months.
  Interventions: Drug: Cidan capsule
- Control group (No Intervention): Patients were only accepted operation and TACE.

INTERVENTIONS:
Drug: Cidan capsule
  Arms: Cidan capsule

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignances seen in different regions of the world. The 5-year risk of recurrence of HCC after resection has been reported to be as high as 70%. It has been proposed that best way to reduce recurrence is to search for improved adjuvant therapies. Especially for some postoperative patients who were identified with the risk factors for recurrence, several adjuvant therapies were often used, including TACE. Recently, a variety of Traditional Chinese Medicine combined with TACE for toxicity reduction and enhancing the efficacy have been investigated in the treatment of HCC. Cidan capsules are a formula containing more than ten types of plant extracts, and has been clinically used for >10 years as a safe and nontoxic antitumor drug. However, the safy and efficacy of preventive therapy is still not clear. In this prospective control study, we enroll such HCC patients experienced operation and were identifed with high risk of recurrence. After a preventive TACE, the eligible patients were divided into two groups. One group will accept Cidan therapy and another will not. Under a basis of large sample, the safty and efficacy of Cidan combined with TACE in HCC patients will be investigated and analysed.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignances seen in different regions of the world. Surgical resection provides the best chance of cure for selected patients. However, we have long been perplexed by high rates of tumor recurrence, which is often the main cause of long-term treatment failure. The 5-year risk of recurrence of HCC after resection has been reported to be as high as 70%. It has been proposed that best way to reduce recurrence is to search for improved adjuvant therapies. Especially for some postoperative patients who were identified with the risk factors for recurrence, several adjuvant therapies were often used, including TACE. However, the safy and efficacy of preventive therapy is still not clear.

Recently, a variety of Traditional Chinese Medicine combined with TACE for toxicity reduction and enhancing the efficacy have been investigated in the treatment of HCC. Cidan capsules are a formula containing more than ten types of plant extracts, including Rhizoma Curcumae (19%), Astragalus (19.6%), Cremastra appendiculata (9.8%), Salvia miltiorrhiza (9.8%), hive (9.8%) and Bombyx batryticatus (9.8%). Cidan has been clinically used for >10 years as a safe and nontoxic antitumor drug. A number of studies have investigated the clinical application of TCMs for HCC, demonstrating that β-elemene, which is present in Rhizoma Curcumae and the main component of cidan, may inhibit the proliferation of HepG2 cells in a time- and dose-dependent manner. The results indicated that β-elemene exhibited positive effects on apoptosis and induced the cell cycle arrest of HepG2 cells in the G2/M phase, while Fas and Fas ligand expression levels were markedly increased.

In this prospective control study, we enroll such HCC patients experienced operation and were identifed with high risk of recurrence. After a preventive TACE, the eligible patients were divided into two groups. One group will accept Cidan therapy and another will not. Under a basis of large sample, the safty and efficacy of Cidan combined with TACE in HCC patients will be investigated and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCC confirmed by pathology.
* Liver function of Child-Pugh Class A or B.
* no intrahepatic and extrahepatic metastasis.
* Tumors had not invaded the portal vein, the hepatic vein trunk or the secondary branches.
* Patients undergone operation were confirmed to have the following high-risk recurrence factors:

Satellite nodules, Poor differentiation, Tumor diameter > 5cm

* No evidence of coagulopathy: platelet count > 50 × 109/L and a prolonged prothrombin time of < 5 seconds.
* The patients would like to accept postoperative TACE.

Exclusion Criteria:

* Informed consent not available
* Impaired liver function with either clinically detected ascites, hepatic encephalopathy, serum albumin < 25g/L or bilirubin > 50micromol/L
* Renal impairment with creatinine > 200micromol/L
* Severe concurrent medical illness persisting > 6 weeks after hepatectomy
* History of other cancer
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Recurrence-free survival | 3 years

OTHER OUTCOMES:
Number of participants with adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mengchao Wu, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China

REFERENCES:
- [Derived] Zheng DH, Yang JM, Wu JX, Cheng SQ, Zhang SG, Wu D, Li AJ, Fu XH, Li X, Qi FC, Duan WH, Chen JH, Yang ZY, Liang L, Zeng JX, Zheng WD, Wu MC. Cidan Capsule in Combination with Adjuvant Transarterial Chemoembolization Reduces Recurrence Rate after Curative Resection of Hepatocellular Carcinoma: A Multicenter, Randomized Controlled Trial. Chin J Integr Med. 2023 Jan;29(1):3-9. doi: 10.1007/s11655-022-3537-4. Epub 2022 Aug 1. PMID 35915317